CLINICAL TRIAL: NCT01526291
Title: Patient-Reported Outcomes With LASIK:PROWL-1
Acronym: PROWL-1
Status: Completed | Type: Observational
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2010.0103
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Laser in Situ Keratomileusis
Keywords: Myopia; Hyperopia; Astigmatism; Patient-reported outcomes; Patient satisfaction; Refractive Error; Emmetropia; Dry eyes; glare; halos; patient expectations
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Patient Satisfaction; Refractive Errors; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study evaluates a questionnaire designed to measure satisfaction and ophthalmic-related quality of life (QOL)in up to 550 active duty subjects prior to and six months following state-of-the-art laser in situ keratomileusis (LASIK).

DETAILED DESCRIPTION:
The LASIK Quality of Life Collaboration Project (LQOLCP) is a government partnership among the FDA, the Department of Defense, and the National Eye Institute (NEI). This project examines patient-reported outcomes (PROs) following LASIK. This three-phased project is part of FDA's ongoing effort to better monitor and improve the safety and effectiveness of lasers used in LASIK surgery. PROWL-1 is the second phase of the larger LQOLCP project. This prospective, questionnaire-based study will be conducted by the Navy Refractive Surgery Center San Diego in collaboration with the U.S. Food and Drug Administration's (FDA's) Center for Devices and Radiological Health (CDRH) and the National Eye Institute (NEI). The primary purpose of this study is to explore the psychometric properties of a newly developed questionnaire assessing satisfaction and ophthalmic-related quality of life (QOL) in 550 active duty patients over a period of six months prior to and following state-of-the-art laser in situ keratomileusis (LASIK). Specific topics of interest include: functional limitations, dry eye symptoms, pre-operative expectations, depression, anxiety, post-operative symptoms, dispositional optimism, and satisfaction. Additionally, standard-of-care, non-invasive clinical data will be collected pre- and postoperatively (e.g., best corrected visual acuity, manifest refraction, wavefront aberrometry, corneal topography, and other clinical assessments), and analyzed. The questionnaire in this study is a newly developed instrument which, once psychometrically evaluated in this U.S. Navy/FDA/NEI collaboration, will be used in future large-scale, multicenter FDA clinical studies that include civilian refractive surgery centers throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or female active duty service member, of any race, and at least 21 years old at the time of the pre-operative examination.
* Speak and read English fluently, and have the ability to give informed consent.
* Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50 D for myopes or 0.75D for hyperopes during the 12-month period immediately preceding the baseline pre-operative examination.
* Soft contact lens users must have removed their lenses at least 1 week before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses must have removed their lenses at least 4 weeks prior to baseline measurements, and have 2 central keratometry readings and 2 manifest refractions taken at least 1 week apart that do not differ by more than 0.50D in either meridian; mires shall be regular.
* Express strong motivation and potential ability to return for all follow-up examinations through the 6-month follow-up exam under the care of the treating investigator, and have access to transportation to meet follow-up requirements.
* Reside in the greater San Diego, California metropolitan area.
* Have been determined to be a good candidate for the LASIK procedure based on the investigator's assessment of medical ophthalmic health, general cognitive function, and physical and social limitations.
* Have a treatment target of bilateral emmetropia or possibly slight hyperopia (+0.25D).
* Have access to a computer with internet service.
* Consent of the subject's command to participate in the study.

Exclusion Criteria:

* Previous introcular or corneal surgery of any kind in either eye, including any type of surgery for either refractive or therapeutic purposes.
* Female subjects who are pregnant or breast-feeding, or intend to become pregnant during the 6 month duration of the study.
* Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and sumatriptin (Imitrex) or any other tryptan.
* Active ophthalmic disease, neovascularization of the cornea within 1 mm of the intended ablation zone, clinically significant lens opacity, or clinically significant dry eye syndrome unresolved by treatment.
* Evidence of glaucoma or intraocular pressure greater than 22mmHg at baseline.
* Evidence of keratonconus, corneal irregularity, or abnormal videokeratography in either eye.
* Corneal thickness insufficient to allow the residual remaining stromal bed to be no less than 300 microns in each eye. The residual stromal bed thickness will be determined by subtracting both the LASIK flap thickness and depth of the ablation from the total central corneal thickness measured by pachymetry.
* History of recurrent erosions or epithelial basement dystrophy.
* Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active duty service members residing in San Diego, CA and planning to undergo refractive surgery using LASIK for myopia, hyperopia, or astigmatism
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2011-08

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Hofmeister, MD, Principal Investigator — US Naval Medical Center, San Diego; Malvina Eydelman, Principal Investigator — US FDA
Locations (1):
- US Naval Medical Center, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Eydelman M, Hilmantel G, Tarver ME, Hofmeister EM, May J, Hammel K, Hays RD, Ferris F 3rd. Symptoms and Satisfaction of Patients in the Patient-Reported Outcomes With Laser In Situ Keratomileusis (PROWL) Studies. JAMA Ophthalmol. 2017 Jan 1;135(1):13-22. doi: 10.1001/jamaophthalmol.2016.4587. PMID 27893066
- [Result] Hays RD, Tarver ME, Spritzer KL, Reise S, Hilmantel G, Hofmeister EM, Hammel K, May J, Ferris F 3rd, Eydelman M. Assessment of the Psychometric Properties of a Questionnaire Assessing Patient-Reported Outcomes With Laser In Situ Keratomileusis (PROWL). JAMA Ophthalmol. 2017 Jan 1;135(1):3-12. doi: 10.1001/jamaophthalmol.2016.4597. PMID 27893063